CLINICAL TRIAL: NCT00495014
Title: A Single-Blind, Randomized, Placebo-Controlled, Ascending Single Dose and Repeat Dose Study With Once Daily Dosing To Evaluate the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of GSK376501 in Healthy Overweight and Obese Subjects
Brief Title: Study To Investigate The Safety And Metabolism Of GSK376501 In Overweight Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Study Director, GSK
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: DIX109981
Record Dates: First submitted 2007-06-28; First posted 2007-07-02 (Estimated); Last update posted 2010-10-15 (Estimated); Status verified 2010-10

CONDITIONS: Type 2 Diabetes Mellitus
Keywords: GSK376501,; Single Dose,; Dose Escalation,; Healthy Overweight/Obese Volunteer
MeSH Terms: conditions — Diabetes Mellitus, Type 2

INTERVENTIONS:
Drug: GSK376501
Drug: Placebo
  Other Names: GSK376501

SUMMARY:
This study represents the second Phase 1 study with GSK376501 and the goal is to further evaluate its safety and tolerability. The way the human body processes GSK376501 will also be determined.

ELIGIBILITY:
Inclusion Criteria:

* The subject is healthy and overweight/obese, defined as having a body mass index greater than 25 but less than 35kg/m2, inclusive.
* The subject is an adult male or a female of non-childbearing potential between the age of 18 and 65 years, inclusive, at the time of signing informed consent.
* The subject and their partner are willing to use double-barrier method of contraception from the first day of study drug administration until 5 half-lives of the drug have elapsed following the last day of study drug administration.
* The subject demonstrates an ECG with values within ranges specified in the protocol at screening or baseline.
* The subject is capable of giving written informed consent, which includes the ability to read, comprehend and comply with the protocol requirements and restrictions as described in the consent form.

Exclusion Criteria:

* Has a known immediate or delayed hypersensitivity reaction or idiosyncrasy to any medication that is chemically related to the study drug or a history of drug or other allergy that, in the opinion of the physician responsible, contraindicates their participation in the study.
* Has a known allergy to any of the tablet formulation excipients of GSK376501 or pioglitazone (as applicable).
* Has sensitivity to heparin or history of heparin-induced thrombocytopenia.
* Has a history of alcohol abuse or dependence within 12 months prior to the study.
* Has a positive alcohol test at screening or baseline and/or is unwilling to abstain from alcohol for 72 hours prior to the start of dosing until discharged from the clinic and for 72 hours prior to the follow-up visit.
* Is unwilling to abstain from caffeine- or xanthine-containing products for 24 hours prior to each dose and throughout each in-house period, and for 24 hours prior to the follow-up visit.
* The subject smokes or has used tobacco or nicotine-containing products within the 6 months prior to the study, or is positive for urine cotinine at screening or at baseline.
* Is unwilling to refrain from the use of tobacco or illicit drugs during the trial, and/or tests positive for urine cotinine or drugs of abuse at screening or at baseline. At minimum, the list of drugs or classes of drugs that will be screened for include the following: amphetamines, barbiturates, benzoylecgonine, benzodiazepines, cannabinoids, cotinine, and opiates.
* Where participation in the study would result in donation of blood in excess of 500 ml within a 56 day period.
* Has a systolic blood pressure outside the range of 140 to 90mmHg, a diastolic blood pressure outside the range of 90 to 60mmHg and/or a heart rate outside the range of 90 to 45bpm, inclusive, at screening or at baseline.
* Experiencing clinically significant ECG abnormalities at screening or at baseline.
* Has a history or current evidence of a positive HIV test.
* Has a history of or a positive pre-study Hepatitis B surface antigen or positive Hepatitis C antibody result within 3 months of screening.
* Has laboratory safety screening tests outside of ranges specified in the protocol at screening or at baseline. T.
* Pregnant or lactating women, or woman of childbearing potential.
* Has a history of rhabdomyolysis.
* Has congestive heart failure or a history of congestive heart failure with New York Heart Association Class I-IV symptoms
* Has a history of thyroid dysfunction or an abnormal thyroid function test as assessed by TSH at screening.
* Has a history or current evidence of sleep apnea.
* Has had previous exposure to GSK376501, with the exception of subjects randomized into a previously completed study with GSK376501 may participate only in the cohort evaluating pioglitazone.
* Has had treatment with any other new molecular entity (investigational drug) during the previous 30 days or 5 half-lives, or twice the duration of the biological effect of the drug (whichever is longer), prior to the first dose of current study medication. For the purposes of this study, a new molecular entity is defined as any compound that has not yet reached Phase 3 development. The washout is defined from last dose of study medication in the previous study until the first dose of study drug.
* Has been exposed to more than four new molecular entities within 12 months prior to the first dosing day.
* Has used the following prescription or non-prescription medications within 14 days or 5 half lives, whichever is longer, prior to the first dose of study medication: vitamins (at a dose greater than the recommended daily allowance), or dietary or herbal supplements, including St. John's Wort.
* Is unable or unwilling to discontinue use of acetaminophen 72 hours prior to each dose and throughout each in-house period and no use within 72 hours of the follow-up visit.
* Requires the use of a prohibited medication .
* Is unable or unwilling to abstain from the consumption of grapefruit or grapefruit juice for 7 days prior to the first dose of study medication until the final pharmacokinetic sample has been collected.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2007-06; Primary Completion 2007-12 (Actual); Study Completion 2007-12 (Actual)

PRIMARY OUTCOMES:
Adverse reactions and changes in laboratory values, vital signs, and/or ECGs following each dose | following each dose

SECONDARY OUTCOMES:
Blood levels of GSK376501 following 1 day (Part A) or 14 days (Part B) of dosing | following 1 day (Part A) or 14 days (Part B) of dosing
GSK376501 plasma levels to derive pharmacokinetic parameters following single and repeat doses for 14 days
Standard markers that may serve as possible surrogates of volume expansions with GSK376501.
Body weight following 14 days of repeat dosing with GSK376501.

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, MD, MPH, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Evansville, Indiana, United States